CLINICAL TRIAL: NCT04638478
Title: PREselection of Patients at Risk for COgnitive DEcline After Radiotherapy Using Advanced MRI
Status: Recruiting | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Maastricht University Medical Center (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Other Study IDs: PRECODE-MRI
Record Dates: First submitted 2020-11-05; First posted 2020-11-20 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Meningioma
Keywords: Meningioma; Radiotherapy; MRI; Neurocognition
MeSH Terms: conditions — Meningioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: PRECODE-MRI — Patients with meningioma WHO I tumours treated with radiotherapy will be included, undergoing extensive cognitive testing combined with advanced brain MRI scans just before, 3 and 24 months after radiotherapy

SUMMARY:
Meningioma are slow growing and frequently occurring intracranial tumors, responsible for 33% of all asymptomatic intracranial tumors and 13-26% of all symptomatic primary brain tumors. The 10-year survival rate is 72%. A variety of treatment options is available for symptomatic meningioma including surgical removal with or without radiotherapy or radiotherapy alone. These therapies can have negative impact on cerebral functioning.

After high dose radiotherapy for primary or metastatic brain tumors 50-90% of > 6 months' survivors develop irreversible disabling cognitive decline leading to premature loss of independence, reduced Quality of Life (QOL) as well as significant economic burden both at the individual as societal level. Especially for patients with a good prognosis like benign meningioma, maintaining neurocognitive function is crucial. Understanding the mechanisms underlying radiation induced cognitive decline is complex and which brain areas to spare are an important subject of research.

Evaluation methods to assess cognitive function and predict cognitive decline are urgently needed, this will allow the development of optimized treatment strategies with the aim to preserve or even improve cognitive function in meningioma patients. Improvements in the field of neuroimaging techniques (i.e. advanced MRI techniques) have the possibility to identify areas susceptible to cognitive impairment. This allows in the future a more personalized radiation treatment by identifying patients at risk, by optimizing the radiotherapy dose to specific brain regions, that could eventually reduce or prevent, cognitive decline. Improvements in the field of radiotherapy for example by higher precision treatment such proton therapy have potential in obtaining these more individualized strategies.

ELIGIBILITY:
Inclusion Criteria:

* Meningioma WHO I, grading based on pathology or radiological features
* Age ≥ 18 years.
* Karnofsky Performance Score 70 or above.
* Ability to comply with the protocol, including neuropsychological testing and imaging.
* Ability to understand the requirements of the study and to give written informed consent, as determined by the treating physician.
* Written informed consent.

Exclusion Criteria:

* Resection meningioma < 3mnd
* Age < 18 years
* Pregnancy
* Any prior cranial radiotherapy
* Any prior chemotherapy in the last 5 years
* Contra-indication for MR imaging (i.e. metal implants, claustrophobia)
* Any other serious medical condition that could interfere with follow-up.
* Severe aphasia or language barrier interfering with assessing endpoints (i.e. completion of questionnaires or neurocognitive performance)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (18 years or older) patients with meningioma tumours (WHO I) in a good clinical condition treated with curative intend using radiotherapy (proton or photon) without other known malignancies.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Estimated)
Dates: Start 2021-04-08 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Correlation cognitive failure and radiotherapy dose | 2 years after radiotherapy
  Correlation between the delta cognitive failure score (baseline vs 2 years) and radiotherapy dose in cognition related brain regions (supratentorial brain, hippocampus left/right and anterior/posterior, cerebellum anterior/posterior).

SECONDARY OUTCOMES:
Correlation baseline imaging and patient specific parameters | 2 years after radiotherapy
  Correlation between baseline imaging (advanced MRI sequence) and patient specific parameters (e.g. baseline cognitive status, age, Karnofsky index (KPS), co-morbidity, alcohol consumption, smoking, medication)
RT induced cognitive change measured with extensive cognitive testing | 2 years after radiotherapy
  RT-induced cognitive change measured with extensive cognitive testing
Correlation advanced MRI and PROMS | 2 years after radiotherapy
  Correlation of advanced MRI and treatment/dose parameters to PROMS; EQ/5D, QLQ/C30, QLQ/BN20, Cognitive Failure questionnaire (CFQ) , Multidimentional Fatigue Index (MVI/20)
Radiation susceptibility of organs by Normal Tissue Complication Probability (NTCP) | 2 years after radiotherapy
  Identification of radiation susceptibility of individual anatomical and functional central nervous system (CNS) organs (e.g. (hippocampi, frontal lobe, cerebellum, brain) for radiation damage by relating dose-volume histogram of the organs with information with neurocognitive test results.
Sensitivity neurocognitive tests | 2 years after radiotherapy
  Sensitivity of additional extensive neurocognitive tests
Correlation advanced MRI and radiotherapy modality | 2 years after radiotherapy
  Correlation of advanced MRI and treatment/dose parameters and radiotherapy modality (photon vs proton)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Zegers, Study Chair — Maastro Clinic, The Netherlands; Danielle Eekers, Principal Investigator — Maastro Clinic, The Netherlands
Locations (1):
- Maastricht Radiation Oncology, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No